CLINICAL TRIAL: NCT02178761
Title: Comprehensive Imaging and Interventional Therapy Studies for Arteriogenic Erectile Dysfunction and Lower Urinary Tract Symptoms: A Multi-modality, Multi-Specialty Collaborative Study (PERFECT Program)
Brief Title: Imaging and Interventional Study for Erectile Dysfunction and Lower Urinary Tract Symptoms
Acronym: PERFECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201402003RINA
Record Dates: First submitted 2014-06-22; First posted 2014-07-01 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Erectile Dysfunction; Lower Urinary Tract Symptoms; Peripheral Arterial Disease
Keywords: Erectile dysfunction; Lower Urinary Tract Symptoms; Peripheral Arterial Disease; Angioplasty; Multidetector Computed Tomography
MeSH Terms: conditions — Erectile Dysfunction; Lower Urinary Tract Symptoms; Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Angioplasty alone (Active Comparator): plain old balloon angioplasty alone
  Interventions: Device: Apex™ PTCA Dilatation Catheter
- Stenting (Active Comparator): Balloon angioplasty plus stenting
  Interventions: Device: Stent System
- drug-eluting balloon (Active Comparator): Balloon angioplasty with drug-eluting balloon
  Interventions: Device: drug-eluting balloon
- biodegradable vascular scaffold stent (Active Comparator): Stenting with biodegradable vascular scaffold stent
  Interventions: Device: biodegradable vascular scaffold stent

INTERVENTIONS:
Device: drug-eluting balloon — angioplasty completed with drug-eluting balloons
  Other Names: SeQuent® Please
  Arms: drug-eluting balloon
Device: biodegradable vascular scaffold stent — Stenting with biodegradable vascular scaffold stents
  Other Names: Absorb Bioresorbable Vascular Scaffold System
  Arms: biodegradable vascular scaffold stent
Device: Apex™ PTCA Dilatation Catheter — plain old balloon angioplasty alone
  Other Names: TREK & MINI TREK Coronary Dilatation Catheter; Sprinter Legend RX
  Arms: Angioplasty alone
Device: Stent System — stenting with either bare-metal stents or drug-eluting stents
  Other Names: Promus PREMIER™ Everolimus-Eluting Platinum Chromium Coronary Stent System; XIENCE PRIME Everolimus Eluting Coronary Stent System; Resolute Integrity Coronary Stent System; BioMatrix Flex™; Nobori® Drug Eluting Stent; MULTI-LINK 8 Coronary Stent System; Integrity Coronary Stent System
  Arms: Stenting

SUMMARY:
Erectile dysfunction is highly prevalent as men grow older. Among the various causes of erectile dysfunction, it has been shown that pelvic arterial insufficiency plays a very important role. The investigators have recently developed the first imaging analytical algorithm by using the abdominal/pelvis multidetector computed tomographic (MDCT) angiography to delineate the whole arterial system supplying the penis. To establish a comprehensive, cutting-edge diagnostic and interventional therapeutic program for erectile dysfunction, the investigators therefore design this series of studies by including experts from Urology, Radiology, and Cardiology. This research project (PERFECT program) includes the following 4 sub-studies: 1) differential frequency of obstructive pelvic arterial lesions in coronary artery disease patients with and without erectile dysfunction/lower urinary tract symptoms (LUTS), 2) differential frequency of obstructive pelvic arterial lesions in patients with vascular risk factors and with or without erectile dysfunction/LUTS, 3) safety, feasibility, and efficacy of comprehensive pelvic angioplasty (with various interventional strategies/instruments) for patients with erectile dysfunction/LUTS and pelvic obstructive arterial disease: proof-of-concept study; and 4) efficacy and safety of comprehensive pelvic angioplasty (with various interventional strategies/instruments) for patients with erectile dysfunction/LUTS and pelvic obstructive arterial disease: a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* men 20 years of age or older with "consistent" erectile dysfunction defined as both IIEF-5 scores, taken at least 4 weeks apart, are in the range of 5 to 21 points and with a difference of <=2 points
* the anatomical inclusion criteria, based on pelvic CT angiography, are unilateral luminal diameter stenosis >=70% or bilateral diameter stenoses >=50% in the pelvic arteries with reference vessel diameter >=2.5 mm and <=4.0 mm and a target-lesion length <=40 mm

Exclusion Criteria:

* the arterial inflow to the penis is entirely from the accessory pudendal arteries rather than the usual internal pudendal artery and common penile artery;
* the presence of focal diameter stenosis >=70% in the common iliac artery, internal iliac artery, or anterior division of internal iliac artery;
* previous radical prostatectomy, pelvic radiation, or Peyronie's disease;
* untreated hypogonadism (serum total testosterone <300 ng/dL within 14 days before enrollment);
* acute coronary syndrome, stroke, or life-threatening arrhythmia within 3 months before enrollment;
* poorly controlled diabetes mellitus with glycosylated hemoglobin levels >9%;
* serum creatinine levels >2.5 mg/dL;
* bleeding diathesis or known hypercoagulopathy;
* life expectancy of fewer than 12 months;
* known intolerance to contrast agents

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-10; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
IIEF | 1 year
  IIEF: Internal index for erectile function
EPS | 1 year
  EPS: erectile hardness score
IPSS | 1 year
  IPSS: international prostate symptom score

SECONDARY OUTCOMES:
CT angiographic binary restenosis | 1 year
  CT angiographic binary restenosis: ≥50% lumen diameter stenosis

OTHER OUTCOMES:
Any major adverse events | 1year

CONTACTS AND LOCATIONS:
Overall Officials: Tzung-Dau Wang, MD, PhD, Principal Investigator — NTUH
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Wang TD, Lee WJ, Yang SC, Lin PC, Tai HC, Hsieh JT, Liu SP, Huang CH, Chen WJ, Chen MF. Safety and six-month durability of angioplasty for isolated penile artery stenoses in patients with erectile dysfunction: a first-in-man study. EuroIntervention. 2014 May;10(1):147-56. doi: 10.4244/EIJV10I1A23. PMID 24832642